CLINICAL TRIAL: NCT07178353
Title: Changes in Muscle Mass, Strength, and Muscle Protein Synthesis in Response to 5 Days of Bedrest in Young, Healthy Adults
Brief Title: Human Skeletal Muscle Response to 5 Days of Bedrest in Young Adults
Acronym: FABRIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Chris McGlory, PhD, Associate Professor, Kingston Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6043735
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Muscular Atrophy; Insulin Resistance; Muscle Protein Synthesis
Keywords: magnetic resonance imaging; muscle protein syntheis; muscle disuse atrophy; bedrest; skeletal muscle; insulin sensitivity
MeSH Terms: conditions — Muscular Atrophy; Insulin Resistance; Muscular Disorders, Atrophic | interventions — Bed Rest

STUDY DESIGN:
Intervention Model Description: This study uses a within-subjects, repeated measures design. Single-arm study. Participants will complete a 5-day free-living, baseline testing period, before undergoing 5 days of strict horizontal bedrest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Bedrest (Experimental): 19 day study period, consisting of baseline testing, 5 days of free-living (habitual daily activities) immediately followed by 5 days of strict bedrest. Diet controlled and physical activity monitored for entire study period.
  Interventions: Other: Bedrest

INTERVENTIONS:
Other: Bedrest — 5 days of strict bedrest. Participants are allowed to sit up in bed, but will perform any bathing or bathroom activities in a wheelchair.
  Other Names: Horizontal Bedrest

SUMMARY:
The goal of this intervention trial is to characterize skeletal muscle atrophy in healthy, young adults during short term bedrest. The main questions it aims to answer are:

How much do skeletal muscle volume, strength, and fatigue resistance decline during bedrest? How much does whole-body insulin sensitivity change during bedrest? How do mitochondrial function and protein synthesis change during bedrest?

Participants will undergo the following tests before and after a free-living control period and before and after a 5 day period of strict horizontal bedrest:

* Magnetic resonance imaging of the thigh muscles
* Strength testing of the thigh muscles
* Insulin sensitivity testing in response to a mixed meal
* Exogenous glucose oxidation in response to a mixed meal
* Muscle biopsies from the thigh muscles
* Blood samples

DETAILED DESCRIPTION:
Skeletal muscle plays a critical role in physical function and metabolic health, with its maintenance driven by the balance between muscle protein synthesis (MPS) and muscle protein breakdown (MPB). During periods of disuse, such as illness or injury, MPS declines while MPB remains relatively unchanged, leading to muscle loss and atrophy. Short-term disuse, such as bedrest, is commonly experienced through hospitalization, and can result in rapid declines in muscle mass and strength, typically affecting the lower limbs to a greater extent. At the molecular level, bed rest significantly reduces MPS, with durations as little as 3 days showing drastic impairment in skeletal muscle turnover. Additionally, short-term periods of disuse have shown to blunt mitochondrial respiration, affecting the ability for skeletal muscle to produce energy for proper funcitoning and metabolic processes. Diminished skeletal muscle metabolic function directly impacts whole-body metabolic health. Periods of bedrest between 5 and 7 days have shown to decrease whole-body glucose tolerance, increase insulin resistance, and decrease insulin-stimulated leg glucose uptake. All together, these contribute to decreased skeletal muscle mass and strength, and diminished metabolic function, contributing to a decline in overall physical function, health, and well-being. Current studies on short-term bed rest (ex. 5 days) in young adults are limited, and existing research has focused on simulated microgravity models rather than horizontal bed rest, which better represents clinical scenarios. Additionally, no study to our knowledge has explored how the molecular mechanisms that drive MPS change over the course of a 5-day bedrest period. This highlights a need to explore if there are differences in the attrition of synthesis rates of the different protein pools in skeletal muscle (ex. myofibrillar, sarcoplasmic, and mitochondrial).

The purpose of the present study is to investigate changes in leg muscle mass, strength, and whole-body insulin sensitivity over five days of bed rest, as well as examine the time-course changes in molecular mechanisms underlying skeletal muscle turnover. The investigators hypothesize that, compared to the control period, quadriceps muscle size (volume and cross-sectional area), strength/power/fatigue resistance, and whole-body insulin sensitivity will decrease following bedrest. The investigators hypothesize that these outcomes will be linked to decreases in mitochondrial respiratory function and impaired fractional synthetic rates of muscle proteins.

In this repeated-measures design, participants will undergo a five day baseline control period followed by five days of bed rest to compare changes from bedrest to their own free-living control period.

Findings from this study will help inform future research on the impact of short-term, clinically-relevant, bedrest in young adults and aid in the development of targeted interventions to mitigate declines in muscle mass from occurring from acute bouts of muscle disuse.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-30 years
* BMI between 18.5-28 kg/m2
* Weight stable (within ±2kg for 6 months)
* Generally healthy as assessed by medical and physical activity questionnaires
* recreationally active

Exclusion Criteria:

* a BMI < 18.5 and > 28 kg/m2
* the use of insulin to control blood glucose levels
* a history of any cardiovascular, respiratory, metabolic diseases, neuromuscular or bone-wasting diseases
* the use of any medication that may affect muscle protein turnover (e.g. androgen or anabolic hormone therapy, chemotherapy)
* a (family) history of thrombosis, platelet or coagulation disorders, or antiplatelet therapy and the use of anticoagulant medications
* the presence of any unremoved, or partially removed metals underneath the skin
* a history of head or eye injury involving metal fragments
* have some type of implanted electrical device (such as a cardiac pacemaker or neurostimulator)
* have implanted metal objects as a result of surgery, such as artificial joints, aneurysm clips, metal staples
* are, or may be, pregnant
* are wearing metal braces on their teeth.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Quadriceps muscle volume | Day 0, and 5
  Quadriceps muscle volume will be assessed by magnetic resonance imaging.

SECONDARY OUTCOMES:
Muscle strength | Day -14, -9, and 5
  Knee extensor peak torque will be assessed using dynamometry
Knee extensor power | Day -14, -9, and 5
  Peak isotonic power determined at 30% maximal isometric voluntary contraction torque using a dynamometer
Muscle fatiguability | Day -14, -9, and 5
  Knee extensor fatiguability will be determined by the decrease in isotonic power across 40 contractions at 30% MVC using dynamometry.
Muscle cross-sectional area | Day 0 and 5
  Change in quadriceps muscle cross sectional area measured by magnetic resonance imaging scan.
Muscle protein synthesis | Day -5 to 0, day 0 to 1, day 0 to 3, day 0 to 5, day 1 to 3, day 1 to 5, and day 3 to 5.
  Muscle protein synthesis measured as fractional synthesis rate of the myofibrillar, sarcoplasmic, and mitochondrial protein pools within skeletal muscle. These 3 pools will be assessed using combined protocol of skeletal muscle biopsy, stable isotope tracing, cavity ring down spectroscopy with liquid isotope analysis, and gas-chromatography pyrolysis isotope-ratio mass spectrometry.
2-hour plasma glucose incremental area under the curve | Aggregate 2-hour window on day -5, 0, and 5
  Determination of the total rise in plasma glucose during a mixed meal tolerance test, to be assessed by an enzyme-linked immunosorbent assay.
2- hour plasma insulin incremental area under the curve | Aggregate 2-hours on day -5, 0, and 5
  Determination of the total rise in plasma insulin during a mixed meal tolerance test, to be assessed by an enzyme-linked immunosorbent assay.
Postprandial glucose oxidation | Aggregate 3 hours during the mixed meal tolerance test on day -5, 0, and 5
  Measurement of 13C excretion in breath samples using isotope ratio mass spectrometry.
Matsuda Index | 2-hours on day -5, 0, and 5
  Insulin sensitivity measured via the Matsuda Index during a mixed meal tolerance test. Matsuda index values <4.0 indicate insulin resistance, with higher values representing insulin sensitivity.
Mitochondrial Respiratory Function | Day -5, 1, 3, and 5
  Mitochondrial respiration will be assessed using an Oroboros Oxygraph 2000.
Expression of Translational Factors Related to Skeletal Muscle Protein Synthesis | Day 0, 1, 3, and 5
  Activation of translational factors involved in skeletal muscle protein synthesis assessed by western blotting.
Plasma glucose concentration | 2-hour mixed meal tolerance test on day -5, 0, and 5
  Plasma glucose concentration measured during a mixed meal tolerance test.
Serum insulin concentration | 2-hour mixed meal tolerance test on day -5, 0, and 5
  Serum insulin concentration measured during a mixed meal tolerance test
Peak glucose concentration | 2-hour mixed meal tolerance test on day -5, 0, and 5
  Peak glucose concentration measured during a mixed meal tolerance test
Peak insulin concentration | 2-hour mixed meal tolerance test on day -5, 0, and 5
  Peak insulin concentration measured during a mixed meal tolerance test.
Transmission Electron Microscopy Analysis | Day 0, 1, 3, and 5
  Imaging of subsarcolemmal and intermyofibrillar mitochondria to assess change in mitochondrial content from bedrest.
Supine to Stand Test | Day 0, 5
  Orthostatic blood pressure assessment pre and post bedrest, and following recovery after bedrest
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | Day -5, 0, and 5
  Insulin resistance assessed using fasting insulin and glucose levels. Values <1.0 indicate insulin sensitivity, >1.9 and < 2.9 indicates early insulin resistance, and values >2.9 indicate significant insulin resistance

CONTACTS AND LOCATIONS:
Overall Officials: Chris McGlory, PhD., Principal Investigator — Queen's University
Locations (1):
- Queen's Univeristy, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No